CLINICAL TRIAL: NCT04324879
Title: A Open-label, Single-arm, Multicenter Phase Ⅱ Clinical Trial of TQ-B3525 in the Treatment of Relapsed / Refractory Follicular Lymphoma (FL)
Brief Title: A Study of TQ-B3525 in the Treatment of Relapsed / Refractory Follicular Lymphoma (FL)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQ-B3525-II-01
Record Dates: First submitted 2020-03-25; First posted 2020-03-27 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Relapsed / Refractory Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — TQ-B3525

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQ-B3525 tablet (Experimental): TQ-B3525 tablet administered orally.
  Interventions: Drug: TQ-B3525

INTERVENTIONS:
Drug: TQ-B3525 — TQ-B3525 tablet administered 20mg orally, once daily in 28-day cycle.

SUMMARY:
The objective of this study is to evaluate the efficacy of TQ-B3525 in patients with relapsed / refractory follicular lymphoma.

ELIGIBILITY:
Inclusion Criteria:

- 1. Understood and signed an informed consent form. 2. 18 years and older; Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1; Life expectancy ≥ 3 months.

3. Relapsed / refractory FL. 4. At least one measurable lymph node or extranodal lymphoma lesions. 5. Adequate organ system function. 6. Male or female subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 6 months after the last dose of study (such as intrauterine devices , contraceptives or condoms) ；No pregnant or breastfeeding women, and a negative pregnancy test are received within 7 days before the first administration.

Exclusion Criteria:

* 1. Has diagnosed and/or treated additional malignancy within 3 years prior to the first administration.

  2. Has a history of immunodeficiency diseases. 3. Has multiple factors affecting oral medication. 4. Has adverse events caused by previous therapy except alopecia that did not recover to ≤grade 1.

  5. Has received systemic steroid treatment within 7 days before the first administration.

  6. Has received other systemic anti-tumor medications within 4 weeks before the first administration, or still within the 5 half-life of the medication, which occurs first.

  7. Has palliative radiation therapy within 4 weeks before the first administration.

  8. Has received surgery, or unhealed wounds within 4 weeks before the first administration.

  9. Has a history of autologous hematopoietic stem cell transplant within 3 months or allogeneic hematopoietic stem cell transplant within 6 months.

  10.Has cardiovascular disease ≥grade 2 within 6 months before the first administration.

  11. Has active hepatitis B or C. 12. Has psychotropic substances abuse or a mental disorder. 13.Has other conditions that make it inappropriate for the patient to be enrolled based on investigator's opinion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-05-20 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) assessed by Independent Review Committee (IRC) | Baseline up to 18 months
  Percentage of subjects achieving complete response (CR) and partial response (PR) based on IRC.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Baseline up to 18 months
  PFS was defined as the time from the date of study enrollment to the date of the first of the following events, objective disease progression or death due to any cause.
Overall response rate (ORR) assessed by investigator | Baseline up to 18 months
  Percentage of subjects achieving complete response (CR) and partial response (PR) based on investigator.
Disease control rate（DCR） | Baseline up to 18 months
  Percentage of subjects achieving complete response (CR) and partial response (PR) and stable disease (SD).
Overall Survival (OS) | Baseline up to 24 months
  OS defined as the time from the first dose to death from any cause. Survival time was censored at the date of last contact for patients who were still alive or lost to follow-up.
Disease control rate (DOR) | Baseline up to 18 months
  DOR defined as time from earliest date of disease response to earliest date of disease progression based on radiographic assessment.
Safety | Baseline up to 18 months
  AE, ADR, and SAE, and withdrawal from the trial for reasons such as safety or tolerability.
Biomarkers | Baseline up to 18 months
  To assess the changes of genes related to PI3K pathway and bypass in the tissues and / or plasma of enrolled patients.

CONTACTS AND LOCATIONS:
Locations (41):
- China (41):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Luohe Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Shijitan Hospital, Beijing, Beijing Municipality
  - Beijing Tsinghua Chang Gung Hospital, Beijing, Beijing Municipality
  - Chinese People's Liberation Army General Hospital, Beijing, Beijing Municipality
  - Fifth Medical Center of General Hospital of Chinese People's Liberation Army, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - The Sixth Medical Center of General Hospital of Chinese People's Liberation Army, Beijing, Beijing Municipality
  - Xuanwu Hospital of Capital Medical University, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Fujian Provincial Cancer Hospital, Fuzhou, Fujian
  - First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Gansu Cancer Hospital, Lanzhou, Gansu
  - Chinese People's Liberation Army Joint Logistics Support Unit 940 Hospital, Lanzhou, Gansu
  - Foshan First People's Hospital, Foshan, Guangdong
  - Sun-Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Cancer Hospital of Guangxi Medical University, Nanning, Guangxi
  - The First Affiliated Hospital of Hainan Medical College, Haikou, Hainan
  - The Second Affiliated Hospital of Hainan Medical College, Haikou, Hainan
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Jiangsu Provincial Cancer Hospital, Nanjing, Jiangsu
  - Affiliated Zhongshan Hospital of Dalian University, Dalian, Liaoning
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Weifang People's Hospital, Weifang, Shandong
  - Weihai Central Hospital, Weihai, Shandong
  - Tongji Hospital of Tongji University, Shanghai, Shanghai Municipality
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality
  - General Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - First People's Hospital of Yunnan Province, Kunming, Yunnan
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Affiliated to Zhejiang University School of Medicine,Sir Run Run Shaw Hospital, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Wang H, Feng J, Liu Y, Qian Z, Gao D, Ran X, Zhou H, Liu L, Wang B, Fang M, Zhou H, Huang Z, Tao S, Chen Z, Su L, Su H, Yang Y, Xie X, Wu H, Sun P, Hu G, Liang A, Li Z. Phase II study of novel orally PI3Kalpha/delta inhibitor TQ-B3525 in relapsed and/or refractory follicular lymphoma. Signal Transduct Target Ther. 2024 Apr 17;9(1):99. doi: 10.1038/s41392-024-01798-0. PMID 38627366